CLINICAL TRIAL: NCT01481376
Title: Laparoscopic Transabdominal Preperitoneal (TAPP) Inguinal Hernia Repair With Self-fixating Parietex™ ProGrip™ Mesh: A Retrospective Study With 12 Month Follow-up
Brief Title: TAPP Inguinal Hernia Repair With Self-fixating Parietex™ ProGrip™ Mesh
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVPTAP0161
Record Dates: First submitted 2011-10-24; First posted 2011-11-29 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-12

CONDITIONS: Postoperative Complications
Keywords: Parietex™ ProGrip™; Laparoscopic Transabdominal preperitoneal; TAPP; Inguinal hernia repair
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this retrospective study is to evaluate the postoperative clinical outcomes at discharge, 1 month and 12 months, associated with the use of Parietex™ ProGrip™ in Laparoscopic Transabdominal preperitoneal inguinal hernia repair. Results from this study will be used to support the short- and long-term clinical outcomes of Parietex™ ProGrip™ when used in inguinal hernia repair by laparoscopic approach.

* Single center study
* Population: All subjects have undergone Laparoscopic Transabdominal preperitoneal surgical treatment for inguinal hernia repair with Parietex™ ProGrip™ without additional fixation between September 2008 and March 2010 (inclusive) with at least 12 months of follow-up.

The primary outcome:

• Proportion of subjects who experience hernia recurrence (defect treated initially with Parietex™ ProGrip™) within 12 months post-surgery.

Recurrence is defined as a clinically manifest bulge or a protrusion exacerbated by a Valsalva maneuver in the operated groin.

The recurrence symptoms are assessed by phone based on the Symptoms Questionnaire and the recurrence diagnosis is confirmed during a physical examination by a physician and defined as a clinically manifest bulge or a protrusion exacerbated by a Valsalva maneuver in the operated groin. If subject has a surgical repair of the hernia within the 12 month postoperative period, it will be documented as evidence of hernia recurrence.

The secondary outcome:

* Incidence of Groin Pain (pain score 0-10) and analgesic use at discharge, 1 month and 12 month postoperatively
* Incidence of postoperative complications including, wound infection (any infection of the incision), mesh infection (an infection of the mesh), bleeding, mesh migration, mesh erosion, fistula, small bowel obstruction, seroma, hematuria, hematoma, inflammation, chronic pains/ inguinodynia, infection, visceral adherence, allergic reactions to the components of the product at discharge, 1month and 12 month post-operatively
* Patient satisfaction
* Operative time
* Hospital length of stay

ELIGIBILITY:
Inclusion Criteria:

* The following diagnosis will be included:

  * Inguinal hernia: unilateral or bilateral

All subjects must meet the following inclusion criteria:

* ≥18 years of age
* Had undergone elective (non-emergent) primary surgical repair of the above diagnosis with Parietex ProGrip™ by Laparoscopic Transabdominal preperitoneal inguinal hernia repair between September 2008 to March 2010
* Post-operative follow-up ≥ 12 months or recurrence which occurs within the 12 months post-surgery (If subject has a known incidence of recurrence before the 12 months follow up, the subject will be included in the study.)

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria are not eligible for study participation:

  * Patients with previous laparoscopic Inguinal hernia repair
  * Emergency procedures
  * Patients with incarcerated hernias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects have undergone Laparoscopic Transabdominal preperitoneal surgical treatment for inguinal hernia repair with Parietex™ ProGrip™ without additional fixation between September 2008 and March 2010 (inclusive) with at least 12 months of follow-up. Subjects must meet the protocol outlined eligibility criteria to be included in the study.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dieter BIRK, MD, Principal Investigator — Evangelisches Krankenhaus Zweibrücken - Obere Himmelsbergstr. 38 - 66482 Zweibrücken - GERMANY
Locations (1):
- Evangelisches Krankenhaus Zweibrücken - Obere Himmelsbergstr. 38, Zweibrücken, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Parietex Progrip: Surgical cure of inguinal hernia using the Parietex™ ProGrip™ mesh by Laparoscopic Transabdominal Preperitoneal (TAPP) approach
Period: Overall Study
Arm/Group | Parietex Progrip
Started | 200
Completed | 169
Not Completed | 31

BASELINE CHARACTERISTICS:
Arm/Group | Parietex Progrip
Number analyzed (Participants) | 169
Age, Continuous [Mean (Full Range); unit: years] | 54.7 [21 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 156

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Experience Hernia Recurrence (Defect Treated Initially With Parietex™ ProGrip™) Within 12 Months Post-surgery.
Description: Recurrence is defined as a clinically manifest bulge or a protrusion exacerbated by a Valsalva maneuver in the operated groin. The recurrence symptoms are assessed by phone based on the Symptoms Questionnaire and the recurrence diagnosis is confirmed during a physical examination by a physician.
Time Frame: At least 12 months post-surgery
Measure: Number; unit: participants
Arm/Group | Parietex Progrip
Number analyzed (Participants) | 169
participants | 3

2. Secondary Outcome: Incidence of Groin Pain (Pain Score 0-10)
Time Frame: 12 month post-operatively
Measure: Number; unit: participants
Arm/Group | Parietex Progrip
Number analyzed (Participants) | 168
participants
  No/Low Pain (score 0-3) | 160
  Mild pain (Score 4-6) | 6
  Severe (score 7-10) | 2

3. Secondary Outcome: Analgesic Use
Time Frame: The day of the discharge (an expected average of 1 day), 1month and at least 12 month post-operatively
Reporting Status: Not Posted

4. Secondary Outcome: Postoperative Complications Including, Infection, Seroma, Hematoma, Visceral Adherence, Allergy Etc
Time Frame: up to 12 months
Measure: Number; unit: participants
Arm/Group | Parietex Progrip
Number analyzed (Participants) | 169
participants
  Hematoma/Seroma | 3
  Emphysema in the inguinal regions (both sides) | 1
  Secondary hemorrhage through the trocar's site | 2
  Hematuria | 1
  Swelling above the genital organs | 1

5. Secondary Outcome: Patient Satisfaction
Time Frame: at least 12 month post-operatively
Measure: Number; unit: participants
Arm/Group | Parietex Progrip
Number analyzed (Participants) | 169
participants
  Very satisfied/Satisfied | 162
  Neutral | 2
  Unsatisfied/Very unsatisfied | 5

6. Secondary Outcome: Operative Time
Time Frame: From skin incision to closure (The expected median operating time is 36 minutes for unilateral and 50 minutes for bilateral repair)
Reporting Status: Not Posted

7. Secondary Outcome: Hospital Length of Stay
Time Frame: Duration of the hospital stay (expected average of 1 day)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Parietex Progrip
Number analyzed (Participants) | 169
Days | 2.1 (0.8)

ADVERSE EVENTS:
Arm/Group | Parietex Progrip
Serious Adverse Events (participants affected / at risk) | 0/169
Other Adverse Events (participants affected / at risk) | 0/169

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less